CLINICAL TRIAL: NCT03990077
Title: A Phase I , Single Arm, Dose Escalation Study to Evaluate Tolerability, Safety, Pharmacokinetics and Preliminary Efficacy of HL-085 Plus Docetaxel in Patients With KRAS Mutant NSCLC
Brief Title: Study of HL-085 Plus Docetaxel in Patients With KRAS Mutant NSCLC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: drug development strategy adjustment
Sponsor: Shanghai Kechow Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HL-085-103
Record Dates: First submitted 2019-06-12; First posted 2019-06-18 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2020-12

CONDITIONS: Nsclc
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Intervention Model Description: If no Dose-limiting toxicity (DLT) occurs in the first three subjects in Cycle 1, the dose will be escalated to the next dose level; If a DLT occurs in one of the first three subjects, three additional subjects will be enrolled for the same dose cohort, and undergo the same procedures. Dose -escalation is performed based on the scheduled dose groups until DLT occurs in two or more subjects in a dose group which consists of 3 or 6 subjects.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dose escalation of HL-085 plus Docetaxel (Experimental): HL-085 will be administered as BID with specified dose. And Docetaxel will be taken as the instruction in the label ( 75mg/m2，IV).
  f no Dose-limiting toxicity (DLT) occurs in the first three subjects in Cycle 1, the dose will be escalated to the next dose level; If a DLT occurs in one of the first three subjects, three additional subjects will be enrolled for the same dose cohort, and undergo the same procedures. Dose -escalation is performed based on the scheduled dose groups until DLT occurs in two or more subjects in a dose group which consists of 3 or 6 subjects.
  Interventions: Drug: HL-085; Drug: Docetaxel

INTERVENTIONS:
Drug: HL-085 — HL-085 ( Capsule) is one MEK inhibitor.
Drug: Docetaxel — Docetaxel is an antineoplastic drug by inhibiting microtubule depolymerization, and attenuating of the effects of bcl-2 and bcl-xL gene expression.

SUMMARY:
This is a phase I, open label, dose escalation study to evaluate tolerability, safety , pharmacokinetics and efficacy in patients with KRAS mutant NSCLC by using HL-085 and Docetaxel.

ELIGIBILITY:
Inclusion Criteria:

1. KRAS mutation NSCLC.
2. One measurable lesion as defined by RECIST 1.1 criteria for solid tumors.
3. Chemotherapy, immunotherapy or radiotherapy ≥ 4 weeks prior to starting the study treatment.
4. Surgery (except for tumor biopsy) or severe trauma ≤ 14 days prior to starting the study treatment.
5. ECOG performance status of 0-1.
6. Life expectancy ≥ 3 months.
7. Ability to take the medicine orally.
8. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Hypersensitivity to study drug ingredients or their analogues.
2. Prior therapy with MEK-inhibitor.
3. Receiving any other anti-cancer therapy at the same time .
4. Active central nervous system (CNS) lesion.
5. Bleeding symptoms at Grade 3 within 4 weeks prior to starting study treatment.
6. ECG QTcB≥480msec in screening, or history of congenital long QT syndrome；
7. Uncontrolled concomitant diseases or infectious diseases.
8. Retinal diseases (Retinal Vein Occlusion (RVO) or Retinal pigment epithelial detachment (RPED) , et al.).
9. History of HIV,HCV,HBV infection.
10. Interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis will be excluded.
11. Serum HCG test is positive.
12. Other conditions that increase the risk of study and influence the result.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs) | Duration of the study, estimated to be approximately 24 months
  Number of Treatment-Related Adverse Events as Assessed by CTCAE v4.03 will be counted.
Maximum tolerated dose (MTD) | DLTs within the first cycle of therapy (up to 35 days)
  The dose level immediately below the dose level at which more than 2 patients from a cohort of 3 to 6 patients experience a dose-limiting toxicity (DLT)

SECONDARY OUTCOMES:
Overall response rate (ORR) | Duration of the study, estimated to be approximately 24 months
  ORR is the proportion of patients with a best overall response of complete response (CR) or partial response (PR), as assessed per response evaluation criteria in solid tumors (RECIST) v1.1.
Peak Plasma Concentration (Cmax) | Duration of the study, estimated to be approximately 24 months
  Cmax is the maximum plasma concentration of HL-085 or metabolite(s).
Area under the plasma concentration verus time curve(AUC) | Duration of the study, estimated to be approximately 24 months
  AUC of HL-085 or metabolites(s) after repeated dosing

CONTACTS AND LOCATIONS:
Overall Officials: Hongqi Tian, PhD, Study Director — Shanghai Kechow Pharma.
Locations (1):
- Cancer Hospital Chinese Academy of Medical Science, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided